CLINICAL TRIAL: NCT02407392
Title: Acetic Acid Guided Biopsies in Barrett's Surveillance for Neoplasia Detection Versus Non-targeted Biopsies (Seattle Protocol): A Feasibility Study for a Randomised Tandem Endoscopy Trial. The ABBA Study.
Brief Title: "Using Dilute Vinegar to Find Changes in Cells During Endoscopy for Patients With Barrett's Oesophagus" (The ABBA Study)
Acronym: ABBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University Hospitals, Leicester (Other); University of Portsmouth (Other); Brighton and Sussex University Hospitals NHS Trust (Other); Western Sussex Hospitals NHS Trust (Other); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: PHT/2014/73
Record Dates: First submitted 2015-01-27; First posted 2015-04-03 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Acetic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non targeted quadrantic biopsies (Active Comparator): Patients undergo current gold standard Barrett's surveillance with quadrantic Seattle protocol biopsies
  Interventions: Procedure: Non targeted quadrantic biopsies
- Acetic Acid targeted biopsies (Experimental): Patients undergo dye spray gastroscopy with Acetic Acid and targeted biopsies for areas of dysplasia.
  Interventions: Drug: Acetic Acid

INTERVENTIONS:
Drug: Acetic Acid — During endoscopy Acetic acid will be sprayed onto Barrett's oesophagus and targeted biopsies of taken.
  Arms: Acetic Acid targeted biopsies
Procedure: Non targeted quadrantic biopsies — During endoscopy patients will undergo current standard quadrantic Seattle protocol biopsies of Barrett's oesophagus
  Arms: Non targeted quadrantic biopsies

SUMMARY:
Problem statement Barrett's oesophagus is a pre-cancerous condition affecting 375,000 people in the U.K. There is a 0.5-3% yearly risk of progressing to oesophageal cancer, from which only 5% of patients will survive for 5 years after diagnosis. Diagnosing the disease at the stage of dysplasia (pre-cancerous) and early cancer improves survival. This has led to the current surveillance strategy of gastroscopy with non-targeted mapping biopsies taken from the Barrett's oesophagus every two years. The large number of biopsies required is time consuming and expensive, yet dysplasia and cancerous tissue is still missed due to the non-targeted biopsy sampling strategy. Acetic acid has been used effectively in the early detection of cervical dysplasia and cancer, and has also been used with success in a high risk Barrett's population (patients with suspected dysplasia or previously treated dysplasia), but not been studied in the lower risk Barrett's surveillance population. A diagnostic study of non-targeted mapping biopsies (current practice) versus targeted biopsies (acetic acid) in a surveillance population is needed before widespread adoption of this technique is possible.

DETAILED DESCRIPTION:
This is a feasibility study to enable powering of a larger study. The investigators would assume a disease detection of 4.5% with acetic acid chromoendoscopy and 1.5% with protocol driven mapping biopsies. However, these assumptions are largely driven from a single centre cohort study and as such need clarification before they could be used for the purposes of powering a study. Based on the historical cohort studies and wide consultation within the British Society of Gastroenterology research committee and consultation with experts in the field, it is estimated that 200 patients would be reasonable for recruitment to enable the reproducibility and generalisability of this data to be established. The purpose of this study is not to produce statistically significant data in itself but to establish likely event rates and effect size to inform the power calculation for the definitive study.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above
2. Biopsy proven Barrett's metaplasia
3. At least 2cm of Barrett's metaplasia (C0 M2)
4. Willing and able to give informed consent

Exclusion Criteria:

1. Less than 2cm (C0 M2) of Barrett's metaplasia
2. Significant oesophagitis
3. Known or prior oesophageal cancer
4. Known or prior oesophageal dysplasia (indefinite for dysplasia CAN be included)
5. Previous endoscopic therapy
6. Known allergy to acetic acid
7. Previous inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by the ratio of patients approached to recruited, percentage of patients who complete both endoscopies | 18 months
  To determine the feasibility of recruiting 200 Barrett's surveillance patients in 18 months. Ratio of patients approached to recruited, percentage of patients who complete both endoscopies.

SECONDARY OUTCOMES:
Participant acceptability of trial design | 18 months
  To assess participant acceptability of the study design through quantitative measures related to study procedures and in-depth qualitative feedback. Qualitative feedback through semi-structured telephone interviews. Patients will be asked how acceptable they found having two endoscopies and whether they would be willing to undergo a study of similar design. This will measured by responses based on a telephone interview questionnaire.
Comparison of dysplasia rates as assessed by the number of biopsies in each endoscopy required to detect dysplasia | 18 months
  To identify the degree of difference in dysplasia (pre-cancerous changes) detection rates between acetic acid gastroscopy (targeted biopsies) and standard gastroscopic practice (non-targeted mapping biopsies) to inform the power calculation for a definitive study. Number of biopsies in each endoscopy required to detect dysplasia.
Feasibility of training in Acetic Acid technique | 18 months
  Feasibility of training and implementation of acetic acid guided dysplasia detection technique. Online training module with pre and post training examination. Seminar based training day with further examination thereafter and correlation of scores following the above methods. The endoscopists will be tested on a validated video library pre and post training. A further test will be performed following 3-6 months to assess for drop off in ability. Percentage of correct answers will be calculated for each test
Clinician's acceptability of using Acetic Acid technique | 18 months
  To explore the acceptability to clinicians and patients of the concept of using a targeted biopsy technique for surveillance instead of non-targeted, mapping biopsies. Semi-structured qualitative interview to explore clinician's attitude to the use of acetic acid following training and implementation of the study. Clinician's will be asked via a telephone interview on a scale of how confident they would be to use acetic acid alone in the surveillance of Barrett's without performing non-targeted biopsies. Clinical's attitudes will be assessed pre and post training as well as at the end of the study.
Facilitators and barriers to recruitment | 18 months
  To identify potential facilitators and barriers to recruitment and retention for the definitive trial. Qualitative patient interview for both those enrolled in the study and those who have declined to identify themes that may assist recruitment into a larger study. This will be measured by means of a telephone questionnaire.
Number of adverse events | 18 months
  Monitoring of adverse outcomes to describe adverse events for the two methods. Number of adverse events recorded in total.

CONTACTS AND LOCATIONS:
Overall Officials: Pradeep Bhandari, MBBS, MD, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom